CLINICAL TRIAL: NCT04575519
Title: Phase 2b Randomized Double-blind, Placebo-controlled Trial to Estimate the Potential Efficacy and Safety of Two Repurposed Drugs, Acetylsalicylic Acid and Ibuprofen, for Use as Adjunct Therapy Added to, and Compared With, the Standard WHO-recommended TB Regimen (SMA-TB)
Brief Title: Adjunctive Acetylsalicylic Acid and Ibuprofen for Tuberculosis
Acronym: SMA-TB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: National Center for Tuberculosis and Lung Disease, Tbilisi, Georgia (Other); Perinatal HIV Research Unit of the University of the Witswatersrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMA-TB-001
Record Dates: First submitted 2020-08-05; First posted 2020-10-05 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Tuberculosis, Pulmonary; Tuberculosis, MDR; Tuberculosis Infection
Keywords: Tuberculosis; Host-directed therapies; Infectious diseases; Drug-sensitive tuberculosis; Drug-resistant tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Multidrug-Resistant; Latent Tuberculosis; Tuberculosis; Communicable Diseases | interventions — Control Groups; Aspirin; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Multicentre, phase IIB, placebo controlled, randomized, 3-arm trial in DS and MDR TB patient
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Active Comparator): Standard of Care (SoC) TB treatment + placebo twice daily during first 4 weeks of TB treatment followed by placebo once daily for an additional 4 weeks.
  Interventions: Drug: Control group; Drug: SoC TB
- SoC TB + ASA group (Experimental): Standard of Care (SoC) TB treatment + acetylsalicylic acid 300mg twice daily during first 4 weeks of TB treatment followed by aspirin 300mg once daily for an additional 4 weeks.
  Interventions: Drug: ASA group; Drug: SoC TB
- SoC TB + IBU group (Experimental): Standard of Care (SoC) TB treatment + ibuprofen 400mg twice daily during first 4 weeks of TB treatment followed by ibuprofen 400mg once daily for an additional 4 weeks
  Interventions: Drug: IBU group; Drug: SoC TB

INTERVENTIONS:
Drug: Control group — placebo 2 months treatment: 2 tablets during 4 weeks + 1 tablet during 4 weeks
  Other Names: placebo
  Arms: Control group
Drug: ASA group — Acetylsalicylic acid 2 months treatment: 2 tablets during 4 weeks (600 mg daily) + 1 tablet during 4 weeks (300 mg daily)
  Other Names: Acetylsalicylic acid (ASA)
  Arms: SoC TB + ASA group
Drug: IBU group — Ibuprofen 2 months treatment: 2 tablets during 4 weeks (800 mg daily) + 1 tablet during 4 weeks (400 mg daily)
  Other Names: Ibuprofen (IBU)
  Arms: SoC TB + IBU group
Drug: SoC TB — Standard of Care Tuberculosis treatment
  Other Names: Standard of Care Tuberculosis treatment

SUMMARY:
The purpose of this study is to assess the efficacy and safety of 2 repurposed drugs (acetylsalicylic acid and ibuprofen), for use as adjunct therapy added to, and compared with, the standard of care (SoC) WHO-recommended TB regimen in drug-sensitive (DS) and multi-drug resistant (MDR) TB patients.

DETAILED DESCRIPTION:
If eligible and informed consent obtained, patients will be randomized 1:1:1 into one of the following 3 arms, to receive:

1. Standard of Care (SoC) TB treatment + placebo twice daily during the first 4 weeks of TB treatment followed by placebo once daily for an additional 4 weeks. (control group).
2. SoC TB treatment + acetylsalicylic acid 300mg twice daily during the first 4 weeks of TB treatment followed by acetylsalicylic acid 300mg once daily for an additional 4 weeks.
3. SoC TB treatment + ibuprofen 400mg twice daily during the first 4 weeks of TB treatment followed by ibuprofen 400mg once daily for an additional 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 18- 60 years of age
2. Written informed consent in a language they understand. This includes informed consent to be in the trial and informed consent to collect specimens.
3. Laboratory confirmed pulmonary TB (with or without extrapulmonary involvement) defined as a hard copy of a sputum laboratory result that reports M. tuberculosis (Mtb) detection by a WHO-recommended assay -both rapid molecular assays or mycobacterial culture with subsequent speciation are acceptable as inclusion criteria.
4. Women of childbearing potential (including females <2 years post-menopausal) must have a negative pregnancy test at enrolment.
5. Participants must be willing to have an HIV test done unless there is compelling evidence that the patient is HIV-infected at the time of randomization.

Exclusion Criteria:

1. Has a comorbid condition where treatment with aspirin, ibuprofen or other NSAID is indicated (e.g. cardiovascular disease, rheumatic fever, chronic pain, etc.)
2. People institutionalized (incarceration in jail or prison, or due to chronic mental illness). If incarcerated during the study, participants may be terminated, those incarcerated in the first 8 weeks of follow up will be late exclusions and replaced*. Patients either who are planned to be hospitalized or currently hospitalized whilst treated for MDR TB in a TB hospital or ward may be enrolled.
3. Receipt of multi-drug TB treatment (including rifamycin plus isoniazid preventive treatment regimens) for ≥3 days in the 6 months prior to randomization. Participants who have received ≥3 days of TB preventive treatment in the month prior to TB treatment initiation will also be excluded.
4. Currently Pregnancy/breastfeeding. Women who conceive and are found to be pregnant in the first 4 weeks of the trial will be terminated from the trial and excluded from the analysis.
5. Any of the following laboratory parameters taken prior to randomization:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN);
   * Total bilirubin > 2 x ULN;
   * Neutrophil count ≤ 700 neutrophils /mm3;
   * Platelet count < 50,000 cells / mm3
   * Haemoglobin concentration less than 8 g/dL
   * Serum creatinine concentration more than twice the upper limit of normal
6. Co-treatment in the three months prior to randomization, or planned treatment over the course of the trial follow up with any one of the following agents:

   * anticoagulant therapy
   * immune modulating therapy (cancer treatments, any oral or daily use of inhaled steroids;
   * Antacids or proton pump inhibitors - including self-treatment and prescription
7. History or clinical record of sensitivity, asthma or allergy that could be attributed to NSAIDs
8. Weight < 45kg at baseline.
9. History or clinical record suggestive of any of the following in the past two years:

   * peptic ulcer disease or gastro-intestinal bleeding,
   * coagulopathy or other bleeding disorder,
   * renal disease requiring hospitalization - in addition, any prior record at any time of acute kidney injury will be an exclusion criterion.
   * liver disease requiring further investigation or hospitalization,
   * underlying cardiovascular disease or risk factors for cardiovascular disease.
10. Patients with HIV infection (irrespective of ART status) if:

    * CD4 <350 cells/mm3
    * if on ART, unsuppressed (>200 copies/ml) viral load
    * if not on ART, either in the opinion of the attending doctor or according to local ART guidelines, the patient should initiate ART during the 8-week initial placebo or NSAID treatment phase.
11. Alcohol use: potential participant either self-reports or in the investigator's opinion that the patient drinks more than an average of four units/day over a usual week or is a binge drinker (men: 5 or more drinks; women: consume 4 or more drinks, in about 2 hours).
12. Major co-morbid conditions or any other finding which in the opinion of the investigator would compromise the protocol compliance or significantly influence the interpretation of results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 354 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Time to ≥ 67% sustained reduction in the TB score | Week 8 of follow-up
  Time to ≥ 67% sustained reduction in the TB score over the course of TB treatment
Hazard ratio for time to stable culture conversion (SCC) | 24 weeks of TB treatment
  Hazard ratio for time to stable culture conversion (SCC), at least 2 consecutive negative cultures for M. tuberculosis at least 4 weeks apart during the first 24 weeks of TB treatment.

SECONDARY OUTCOMES:
Hazard ratio for stable culture conversion (SCC) at week 8 and week 16 after treatment start. | At week 8 and week 16
  Difference between each intervention arm and control group
Proportion of patients with improvement or resolution of clinical signs and symptoms at end of treatment (TB score). | At week 24
  Difference between each intervention arm and control group
Proportion of patients with improvement of lung function impairment as change from baseline at week 8, 24 and end of treatment in the 1-second forced expiratory volume (FEV1) expressed as FEV1. | At baseline, week 8 and week 24
  Difference between each intervention arm and control group
Changes in the BCN-SA Radiological Score Value. | At baseline, week 8, week 24 (and month 12 if MDR)
  Change in chest-X ray (measured with the BCN-SA score) using the x-ray taken at baseline as the comparator compared with subsequent x-rays over the course of TB therapy. Difference between each intervention arm and control group. The BCN-SA Radiological Score Value assesses the sum of acute and chronic findings in the chest X-ray. Per each finding, a minimum score of 0 and a maximum score of 8 is recorded. The total score value is calculated by adding all the individual findings score values. Higher values of total score represent a worse outcome.
Number of patients with improvement of Health-related Quality of Life comparing baseline measure with that over the course of therapy. | At week 8, week 24 and for MDR TB patients at the end of treatment
  Difference between each intervention arm and control group

OTHER OUTCOMES:
Safety 1: SAEs participant proportion. | Up to month 6 in DS TB patients and up to month 20 in MDR TB patients
  Proportion of participants with at least one serious adverse events (SAEs) by arm until the end of TB treatment, between each intervention arm and the control group.
Safety 2: SAEs in person time. | Up to week 12
  Serious adverse event (SAEs) rate expressed in person time, starting the day of the first dose of NSAID or placebo until one month (30 days) after the last placebo or NSAID taken, including all adverse events recorded in each arm.
Tolerability 1: permanent discontinuity proportion. | Up to week 8
  The proportion of patients in each arm who either permanently discontinued either placebo, acetylsalicylic acid or ibuprofen.
Tolerability 2: treatment interruption proportion | Up to week 10
  The proportion of patients in each arm who had TB treatment interruption for longer than seven days/doses, prescribed either by a listed investigator, or a non-study physician up to two weeks after scheduled or unscheduled permanent discontinuation of placebo/NSAID

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Vilaplana, MD, PhD, Study Chair — Fundació Institut Germans Trias i Pujol
Locations (3):
- National Center for Tuberculosis and Lung Diseases, Tbilisi, Georgia
- South Africa (2):
  - Perinatal HIV Unit (PHRU)- Chris Hani Baragwanath Hospital, Soweto, Johannesburg
  - PHRU- Matlosana, Tshepong Hospital MDR Unit, Klerksdorp, Matlosana

REFERENCES:
- [Derived] Arias L, Otwombe K, Waja Z, Tukvadze N, Korinteli T, Moloantoa T, Fonseca KL, Pillay N, Seiphetlo T, Ouchi-Vernet D, Siles A, Carabias L, Quinones C, Vashakidze S, Martinson N, Vilaplana C. SMA-TB: study protocol for the phase 2b randomized double-blind, placebo-controlled trial to estimate the potential efficacy and safety of two repurposed drugs, acetylsalicylic acid and ibuprofen, for use as adjunct therapy added to, and compared with, the standard WHO recommended TB regimen. Trials. 2023 Jun 28;24(1):435. doi: 10.1186/s13063-023-07448-0. PMID 37370174
- See also: CORDIS -CE database -SMA-TB project description — https://cordis.europa.eu/project/id/847762
- See also: SMA-TB repository — https://zenodo.org/communities/sma-tb/?page=1&size=20